CLINICAL TRIAL: NCT05391334
Title: Exploration and Comparison of Novel Technology-supported Methods for Early Fall Risk Detection and Fall Prevention Among Inpatients With Delirium
Brief Title: Early Fall Risk Detection and Fall Prevention Among Inpatients With Delirium
Acronym: QumPreFall
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Department of Geriatric Medicine FELIX PLATTER (Other)
Collaborators: University of Basel (Other); Velux Stiftung (Unknown)
Responsible Party: Sponsor
Other Study IDs: QumEKNZV2
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Delirium in Old Age; Delirium Superimposed on Dementia; Fall; Bed Falls
Keywords: bed-exit; bed-exit warning device; contact mat; 3-D-radar device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual Care: Contact mat (CareMat®) for bed-exit detection in combination with Qumea fall detection.
- Intervention: Contactless motion sensor (Qumea®) for bed-exit detection in combination with Qumea fall detection.
  Interventions: Device: Qumea

INTERVENTIONS:
Device: Qumea — Contactless motion sensor (Qumea®) for bed-exit detection in combination with Qumea fall detection.
  Groups: Intervention

SUMMARY:
During delirium patients are at risk of severe harm due to unattended bed-exits resulting in falls. This research intends to explore how effective alarming contact mats (CareMat®) in comparison to contactless bed-exit alarming devices (Qumea®) are to reduce the risk of unattended bed-exits and falls.

DETAILED DESCRIPTION:
Delirium is a neuropsychiatric disorder with a sudden and reversible decline in attention and cognition due to a medical condition.8 Delirium is associated with emotional distress for patients, their relatives and medical staff.3-5 During delirium, patients are at risk of severe harm due to unattended bed-exits and subsequent falls.6, 7 As worldwide strategy, sitters are used for the prevention of harm in patients with delirium. However, evidence of the effectiveness of sitters is scant.9 A newly designed specialised acute care unit for older patients with delirium, the FELIX PLATTER delirium unit (DelirUnit), strives to overcome the aforementioned shortcomings. On the DelirUnit there are no physical barriers such as bed rails to prevent patients from bed-exits. Floor beds minimize injuries when patients leave their beds unattended. Specialised nurses and nursing aides care for this vulnerable patient group. Sitters are banned. As an alternative to sitters, nurses are informed about patients' intended bed-exit by electronic alarming contact mats at the bedside or in front of beds (CareMat®) or by a novel contactless radar-based bed-exit monitoring system (Qumea®). Up until now, evidence for the effectiveness of technical devices for fall risk prevention is low. This research intends to explore how effective contact mats (CareMat®) or contactless bed-exit alarming devices (Qumea®) are in fall risk detection and fall prevention.

ELIGIBILITY:
Inclusion Criteria:

Admission at or transferal to DelirUnit. During Covid pandemic, patients will be enrolled into the study after the second negative Covid swab (PCR).

Exclusion Criteria:

Patients who have been sectioned and must be treated in a facility, whether they agree or not (under the mental health act) (Fürsorgliche Unterbringung).

No proxy consent available due to language barriers;

Missing legal proxy in case of lacking family network

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with delirium hospitalized on a specialized delirium unit
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Falls | 6 months
  Number of patient falls in patient room

SECONDARY OUTCOMES:
Bed-exit patterns | 6 months
  Qumea® provides the following bed-exit pattern categories: 'STANDING', 'SITTING, 'LYING' oder 'OUT_OF_BED' .
  Unit is number/percentage of bed-exit patterns. Artificial intelligence algorithms provide automatized detected bed-exit patterns by a three dimensional radar (Qumea®)
Nurses' workload | 6 months
  Workload is defined as the time in minutes per patient and per day (24-hour period) that a nurse is present in each patient's room. This is measured as the time between activation (nurse enters room) and deactivation (nurse leaves room) of the Hospicall (the hospitals' patient call system) presence button by the nurse in each patient's room. Hospicall automatically generates a time stamp in the logbook of the Hospicall operating system when the presence button is activated and deactivated.
Time to confirm a CareMat® / Qumea® warning by nurse presence in room | 6 months
  Time difference in seconds between timestamps from onset of warning and confirmation of warning with presence button in patient room of bed-exit warning from bed-exit surveillence systems (Qumea® or CareMat®) to Hospicall (a decentralised, scalable patient call system).
  It is the time a nurse needs to confirm a bed-exit warning from the bed-exit surveillence systems.
Delirium severity | 6 months
  Delirium severity is a score between 0 and 39 points on a 13-item 4-point (0-3) Lickert scale, as measured with the Delirium Rating Scale Revised 98 (DRS-R-98). A cut-off score of 15.5 points indicates delirium. The higher the score, the more severe is the delirium. For the prediction models, the DRS-R-98 scores (1) at admission, (2) the mean values of the course of delirium and (3) the difference between admission and discharge will be calculated. The measurements are conducted by the research team (PI or research assistants) during the stay on the delirium unit (on Mondays, Wednesdays and Fridays) and on the day before discharge.
Delirium duration | 6 months
  To determine the duration of delirium, the presence and/or severity of delirium is first measured with the modified Confusion Assessment Method for the Emergency Department (mCAM-ED). The mCAM-ED provides the following categories: (0) no delirium (1) probable delirium (2) definite delirium. Duration of delirium is measured in days between the first delirium positive mCAM-ED assessments (category 1 or 2) and the last delirium positive (category 1 or 2) mCAM-ED assessments. The mCAM-ED assessments are conducted by the research team (PI or research assistants) Mondays, Wednesdays and Fridays and on the day before discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Hasemann, PhD, Principal Investigator — University Department of Geriatric Medicine FELIX PLATTER
Locations (1):
- Universitäre Altersmedizin Felix Platter, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided